CLINICAL TRIAL: NCT02737644
Title: Peri-conception Key Nutritional Factors and Primary Prevention of Congenital Heart Disease(CHD)
Brief Title: Peri-conception Key Nutritional Factors and Congenital Heart Disease
Acronym: PKNFCHD
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Fudan University (Other)
Responsible Party: Sponsor
Other Study IDs: GWIV24_v1
Record Dates: First submitted 2016-04-03; First posted 2016-04-14 (Estimated); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Congenital Heart Disease
Keywords: Congenital Heart Disease; Key Nutritional Factors; conception; pregnant
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- CHD birth cohort: Cases are identified as those whose newborns screened and confirmed with CHD during the follow-up and four age- and delivery-hospital matched controls are selected for each case from the rest of the cohort.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — This is an observational study
  Other Names: This is an observational study

SUMMARY:
The study is a nested case-control study and the purpose is to describe the status of key nutrients(eg.folic acid and vitamins) supplementation among pregnant women in Shanghai, to find out the association between the level of serum key nutrients during peri-conceptional period and the incidence of congenital heart defects (CHD) in newborn, and to provide better preconception care.

DETAILED DESCRIPTION:
Congenital heart defects (CHD) are among the most common major congenital anomalies with an incidence of about 8-12/1,000 live births worldwide. The mechanism of CHD is still unclear. Many studies indicated that the level of key nutrients (eg.folic acid and vitamins) during peri-conceptional period might affect the incidence of CHD, but the evidence is limited. The study aimed to explore the association between serum key nutrients during peri-conceptional period and the incidence of CHD in newborn. All couples attending pre-pregnancy physical examination from 11 districts (Minhang District, Huangpu District, Xuhui District, Changning District, Jingan District, Putuo District, Yangpu District, Jiading District, Pudong District，Songjiang District, Qingpu District) in Shanghai from March 2016, are recruited and their blood samples and questionnaires about the supplementation of key nutrients are collected. During the gestation, venous blood of pregnant women at all of three trimesters is taken. Besides, questionnaires about the supplementation of key nutrients at the first antenatal visit are also obtained. The level of serum folic acid, vitamin A and vitamin B12 at preconception and during gestation are measured. Finally, investigators identifies those whose newborns developed CHD during follow-up as the cases. Then, investigators selects four controls for each case from the rest of the cohort by matching on constitutional determinants of CHD such as age and sex. Participants are identified by national identification number during the follow up. The level of serum key nutrients is compared in cases and controls. Univariate and multivariate association analyses will be performed to identify risk factors to CHD by using multivariate logistic regression model.

ELIGIBILITY:
Inclusion Criteria:

* attend pre-pregnancy physical examination from 11 districts in Shanghai, OR pregnant women present at first antenatal care < 14 week of gestation
* plan to deliver in Shanghai

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All couples attending pre-pregnancy physical examination from 11 districts in Shanghai from March 2016, or pregnant women present at first antenatal care < 14 week of gestation
Sampling Method: Non-Probability Sample
Enrollment: 37000 (Actual)
Dates: Start 2016-03; Primary Completion 2020-12-30 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
preconceptional maternal serum folate level | usually 6 months before pregnancy
  a serum sample collected at preconception and/or early conception will be used for examination

SECONDARY OUTCOMES:
early conceptional maternal serum folate deficiency | first antenatal visit (usually 12th-16th gestational week)
  a serum sample collected at early conception will be used for examination
The status of serum Vitamin D level | periconception period ( defined as around 6 months before and the first 3 months of gestation
  a serum sample collected at preconception and/or first antenatal visit will be used for examination
Pre-conceptional maternal diet folic acid supplement intake | preconception examination (usually 0-6 months before pregnancy)
  a questionnaire administered at preconception and early conception will be used for estimation based on the dose and frequency of supplements intake
Peri-conceptional maternal plasma homocysteine level | peri-conception examination ( defined as about 6 months before and 3 months after conception
  a plasma sample collected at preconception and first antenatal visit will be used for examination
neonatal congenital heart disease(CHD) status | Congenital heart disease screening during 6-72 hours after delivery
  The newborn babies with heart murmurs(≥ 2 grade) and subnormal Pulse Oximetry reading positive will be considered positive-screened and echocardiography will performed.
Peri-conceptional paternal serum folate level | usually between 0-6 months before and 3 months after conception)
  a serum sample collected at preconception and/or early conception will be used for examination

CONTACTS AND LOCATIONS:
Overall Officials: Ying G Huang, PHD, Study Chair — Children's Hospital of Fudan University
Locations (1):
- Children Hospital of Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Reller MD, Strickland MJ, Riehle-Colarusso T, Mahle WT, Correa A. Prevalence of congenital heart defects in metropolitan Atlanta, 1998-2005. J Pediatr. 2008 Dec;153(6):807-13. doi: 10.1016/j.jpeds.2008.05.059. Epub 2008 Jul 26. PMID 18657826
- [Result] Ionescu-Ittu R, Marelli AJ, Mackie AS, Pilote L. Prevalence of severe congenital heart disease after folic acid fortification of grain products: time trend analysis in Quebec, Canada. BMJ. 2009 May 12;338:b1673. doi: 10.1136/bmj.b1673. PMID 19436079
- [Result] Peyvandi S, Rychik J, Zhang X, Shea JA, Goldmuntz E. Preconceptual Folic Acid Use and Recurrence Risk Counseling for Congenital Heart Disease. Congenit Heart Dis. 2015 May-Jun;10(3):219-25. doi: 10.1111/chd.12206. Epub 2014 Jul 24. PMID 25059817
- [Derived] Chen X, Zhang Y, Chen H, Dou Y, Wang Y, He W, Ma X, Sheng W, Yan W, Huang G. Association Between Serum Glycated Hemoglobin Levels at Early Gestation and the Risk of Subsequent Pregnancy Loss in Pregnant Women Without Diabetes Mellitus: Prospective Cohort Study. JMIR Public Health Surveill. 2023 Dec 12;9:e46986. doi: 10.2196/46986. PMID 38085559
- [Derived] Chen H, Zhang Y, Wang D, Chen X, Li M, Huang X, Jiang Y, Dou Y, Wang Y, Ma X, Sheng W, Jia B, Yan W, Huang G; SPCC (Shanghai Preconception Cohort) Group. Periconception Red Blood Cell Folate and Offspring Congenital Heart Disease : Nested Case-Control and Mendelian Randomization Studies. Ann Intern Med. 2022 Sep;175(9):1212-1220. doi: 10.7326/M22-0741. Epub 2022 Aug 23. PMID 35994746
- [Derived] Wang D, Zhang Y, Jiang Y, Ye Y, Ji M, Dou Y, Chen X, Li M, Ma X, Sheng W, Huang G, Yan W; SPCC group. Shanghai Preconception Cohort (SPCC) for the association of periconceptional parental key nutritional factors with health outcomes of children with congenital heart disease: a cohort profile. BMJ Open. 2019 Nov 24;9(11):e031076. doi: 10.1136/bmjopen-2019-031076. PMID 31767586